CLINICAL TRIAL: NCT02998177
Title: Characterization of Rebound Pain Following Peripheral Nerve Block and Its Association With Gut Microbiome Diversity
Status: Completed | Type: Observational
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Dr. David Brenner, Peripheral Nerve Block Fellow, Cork University Hospital
Other Study IDs: GMB-RP
Record Dates: First submitted 2016-11-28; First posted 2016-12-20 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Pain, Postoperative; Gastrointestinal Microbiome
Keywords: Postoperative pain; Rebound pain; Gut microbiome; Gut microbiota; Peripheral nerve block; Axillary brachial plexus block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pre- and postoperative faecal samples and preoperative salivary samples are going to be taken.
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to determine the association between gut microbiome diversity and the characteristics of rebound pain at offset of peripheral nerve block in patients who have undergone upper limb surgery. Other purposes of this study are to determine associations between gut microbiome constitution and persistent post-surgical pain; and describing rebound pain by quantifying its clinical, psychological and neurophysiological characteristics in this patient cohort.

DETAILED DESCRIPTION:
Based on an emerging understanding of the importance of the gut microbiome in the human and animal responses to stress, it is clear that gut microbiota influence bidirectional signaling between the central nervous system (CNS) and gut (microbiota-gut-brain axis). One element of this influence is the role of gut microbiota in visceral hypersensitivity and pain. Important clinical implications of this understanding have begun to emerge: for instance irritable bowel syndrome (IBS) patient cohorts demonstrate distinct gut microbiome characteristics and, in pre-clinical models, manipulation of the gut microbiome lessens visceral hypersensitivity. To date, attempts to improve pain symptoms in IBS using probiotics have been modestly and variably successful.

One research area which offers potential to the discovery of novel analgesic therapies is the activation of endogenous opiate pain processing including augmentation of descending inhibition. (Broadly, identification of new targets/alkaloid modification/ proteomics efforts have been unsuccessful). Manipulation of microbiota-gut-brain axis by administering probiotics offers one potential route for such activation. There are many of examples of such manipulation altering animal behavior and physiology. In theory, opportunities for such manipulation might exist during or close to early life stress or before noxious stimuli such as elective surgery.

The relationship between the gut microbiome and somatic or neuropathic pain has not been studied. Certain of the pathways and regulators of visceral pain and hypersensitivity are also critical in somatic pain handling. These include peripheral sensitization of primary sensory afferents, central sensitization in particular of spinal ascending neurons and alteration of descending inhibitory pathways. These neuroplastic changes have been well documented in the surgical setting in the examination of persistent post-surgical pain.

"Rebound pain" is a quantifiable difference in pain scores when the block is working, versus the increase in acute pain that is encountered during the first few hours after the effects of perineural single-injection or continuous infusion local anesthetics resolve. Rebound pain may represent a manifestation of hypersensitivity and offer an accessible clinical model suitable for examining the association between gut microbiome diversity and perioperative neuroplastic changes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Patients undergoing hand surgery for Dupuytren's contracture correction or open reduction and internal fixation of distal radius fracture under axillary brachial plexus block

Exclusion Criteria:

* Contraindication of regional anaesthesia, patient is allergic to local anesthetics
* Chronic pain syndrome
* History of peripheral neuropathy
* Preexisting nerve damage in the operated arm (sensory or motor deficit)
* Axillary surgery in the past
* Uncontrolled pain (Verbal Rating Score ≥5 out of 10 at rest despite adequate analgesic measures)
* Clinically significant cognitive impairment (Minimental state score < 24)
* Language barrier
* Depression
* Diabetes
* Obesity (BMI>35)
* Antibiotic therapy in the preceding 30 days
* Probiotics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA I-II patients scheduled to undergo upper limb surgery under brachial plexus block will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Association between gut microbiome α diversity and the magnitude of rebound pain (Numerical Rating Scale) | Perioperative period

SECONDARY OUTCOMES:
Association between gut microbiome α diversity and magnitude of postoperative pain (Numerical Rating Scale). | Perioperative period
Association between gut microbiome α diversity and analgesic consumption (mg/24 hours). | Perioperative period
Association between gut microbiome α diversity and salivary cortisol concentration (ng/ml). | Perioperative period
Association between gut microbiome α diversity and Pain Perception Threshold (PPT, mAmp). | Perioperative period
Association between gut microbiome constitution (α diversity) and incidence of persistent post-surgical pain. | Up to 4 weeks postoperatively
Pearson's correlation coefficient for i. Maximum Numerical Rating Scale (NRS) score for rebound pain vs. ii. Pain Perception Threshold (PPT, mAmp) and Pain Tolerance Threshold (PTT, mAmp) based on Quantitative Sensory Testing. | Up to 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: George Shorten, Professor, Study Chair — Professor of Anaesthesia and Intensive Care Medicine, Consultant Anaesthetist, University College Cork / Cork University Hospital
Locations (2):
- Ireland (2):
  - Department of Anaesthesiology, South Infirmary-Victoria University Hospital, Cork, Co. Cork
  - Division of Anaesthesia and Intensive Care, Cork University Hospital, Cork, Co. Cork

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Enck P, Zimmermann K, Menke G, Klosterhalfen S. Randomized controlled treatment trial of irritable bowel syndrome with a probiotic E.-coli preparation (DSM17252) compared to placebo. Z Gastroenterol. 2009 Feb;47(2):209-14. doi: 10.1055/s-2008-1027702. Epub 2009 Feb 5. PMID 19197823
- [Background] Hsiao EY, McBride SW, Hsien S, Sharon G, Hyde ER, McCue T, Codelli JA, Chow J, Reisman SE, Petrosino JF, Patterson PH, Mazmanian SK. Microbiota modulate behavioral and physiological abnormalities associated with neurodevelopmental disorders. Cell. 2013 Dec 19;155(7):1451-63. doi: 10.1016/j.cell.2013.11.024. Epub 2013 Dec 5. PMID 24315484
- [Background] Williams BA, Bottegal MT, Kentor ML, Irrgang JJ, Williams JP. Rebound pain scores as a function of femoral nerve block duration after anterior cruciate ligament reconstruction: retrospective analysis of a prospective, randomized clinical trial. Reg Anesth Pain Med. 2007 May-Jun;32(3):186-92. doi: 10.1016/j.rapm.2006.10.011. PMID 17543812
- [Background] Williams BA. Forecast for perineural analgesia procedures for ambulatory surgery of the knee, foot, and ankle: applying patient-centered paradigm shifts. Int Anesthesiol Clin. 2012 Winter;50(1):126-42. doi: 10.1097/AIA.0b013e31821a00d0. PMID 22227428
- [Background] Clarke SF, Murphy EF, O'Sullivan O, Lucey AJ, Humphreys M, Hogan A, Hayes P, O'Reilly M, Jeffery IB, Wood-Martin R, Kerins DM, Quigley E, Ross RP, O'Toole PW, Molloy MG, Falvey E, Shanahan F, Cotter PD. Exercise and associated dietary extremes impact on gut microbial diversity. Gut. 2014 Dec;63(12):1913-20. doi: 10.1136/gutjnl-2013-306541. Epub 2014 Jun 9. PMID 25021423
- [Background] Lapthorne S, Pereira-Fantini PM, Fouhy F, Wilson G, Thomas SL, Dellios NL, Scurr M, O'Sullivan O, Ross RP, Stanton C, Fitzgerald GF, Cotter PD, Bines JE. Gut microbial diversity is reduced and is associated with colonic inflammation in a piglet model of short bowel syndrome. Gut Microbes. 2013 May-Jun;4(3):212-21. doi: 10.4161/gmic.24372. Epub 2013 Apr 2. PMID 23549027
- [Background] O'Mahony SM, Marchesi JR, Scully P, Codling C, Ceolho AM, Quigley EM, Cryan JF, Dinan TG. Early life stress alters behavior, immunity, and microbiota in rats: implications for irritable bowel syndrome and psychiatric illnesses. Biol Psychiatry. 2009 Feb 1;65(3):263-7. doi: 10.1016/j.biopsych.2008.06.026. Epub 2008 Aug 23. PMID 18723164
- [Background] DuPont AW, DuPont HL. The intestinal microbiota and chronic disorders of the gut. Nat Rev Gastroenterol Hepatol. 2011 Aug 16;8(9):523-31. doi: 10.1038/nrgastro.2011.133. PMID 21844910
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985
- [Background] Melzack R. The McGill pain questionnaire: from description to measurement. Anesthesiology. 2005 Jul;103(1):199-202. doi: 10.1097/00000542-200507000-00028. PMID 15983473
- [Background] Stalder T, Kirschbaum C, Kudielka BM, Adam EK, Pruessner JC, Wust S, Dockray S, Smyth N, Evans P, Hellhammer DH, Miller R, Wetherell MA, Lupien SJ, Clow A. Assessment of the cortisol awakening response: Expert consensus guidelines. Psychoneuroendocrinology. 2016 Jan;63:414-32. doi: 10.1016/j.psyneuen.2015.10.010. Epub 2015 Oct 20. PMID 26563991